CLINICAL TRIAL: NCT05905913
Title: Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of Single- and Multiple-Ascending Doses of Intravenous ANT3310 Alone and in Combination With Meropenem in Healthy Subjects
Brief Title: FiH Study to Assess Safety and PK of SAD and MAD of ANT3310 Alone and in Combination With Meropenem in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Antabio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: ANT3310-1001
Record Dates: First submitted 2023-05-19; First posted 2023-06-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Meropenem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part A: Single Intravenous Ascending Dose of ANT3310 (Experimental)
  Interventions: Drug: ANT3310
- Part A: Single Intravenous Dose of Matching placebo (Placebo Comparator)
  Interventions: Drug: ANT3310-placebo
- Part B: Multiple Intravenous Ascending Doses of ANT3310 (Experimental)
  Interventions: Drug: ANT3310
- Part B: Multiple Intravenous Ascending Doses of Matching Placebo (Placebo Comparator)
  Interventions: Drug: ANT3310-placebo
- Part C: ANT3310 + Meropenem (Experimental): Participants will receive a single intravenous dose of ANT3310 or Meropenem in one of the 2 treatment sequences followed by the repeat administrations of ANT3310 + Meropenem.
  Interventions: Drug: ANT3310; Drug: Meropenem
- Part C: ANT3310 Placebo + Meropenem Placebo (Placebo Comparator): Participants will receive a single dose of ANT3310-placebo or Meropenem-placebo in one of the 2 treatment sequences followed by repeat administrations of ANT3310-placebo + Meropenem-placebo
  Interventions: Drug: ANT3310-placebo; Drug: Meropenem-placebo

INTERVENTIONS:
Drug: ANT3310 — ANT3310 will be infused over 3 hours
  Arms: Part A: Single Intravenous Ascending Dose of ANT3310
Drug: ANT3310-placebo — ANT3310-placebo will be infused over 3 hours
  Arms: Part A: Single Intravenous Dose of Matching placebo
Drug: ANT3310 — ANT3310 will be infused over 3 hours every 8 hours
  Arms: Part B: Multiple Intravenous Ascending Doses of ANT3310
Drug: ANT3310-placebo — ANT3310-placebo will be infused over 3 hours every 8 hours
  Arms: Part B: Multiple Intravenous Ascending Doses of Matching Placebo
Drug: ANT3310-placebo — ANT3310-placebo will be infused over 3 hours as a single dose as part of the drug drug interaction study, then every 8 hours as part of the repeat doses study.
  Arms: Part C: ANT3310 Placebo + Meropenem Placebo
Drug: ANT3310 — ANT3310 will be infused over 3 hours as a single dose as part of the drug-drug interaction study, then every 8 hours as part of the repeat doses study.
  Arms: Part C: ANT3310 + Meropenem
Drug: Meropenem — Meropenem will be infused over 3 hours as a single dose as part of the drug-drug interaction study, then every 8 hours as part of the repeat doses study.
  Arms: Part C: ANT3310 + Meropenem
Drug: Meropenem-placebo — Meropenem-placebo will be infused over 3 hours as a single dose as part of the drug-drug interaction study, then every 8 hours as part of the repeat doses study.
  Arms: Part C: ANT3310 Placebo + Meropenem Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single and multiple intravenous ascending doses of ANT3310, a novel, specific, competitive inhibitor of serine β-lactamases, alone and in combination with meropenem in healthy subjects.

ELIGIBILITY:
Main Inclusion Criteria:

* Participant capable of giving signed informed consent
* Contraceptive use by women or men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Participants are overtly healthy as determined by a medical evaluation including medical history without clinically relevant pathologies, physical examination, vital signs, ECG assessment, and clinical laboratory result
* eGFR ≥ 90 mL/min and < 160 mL/min for males or < 150 mL/min for females
* Body weight within 50.0 and 100.0 kg and BMI within 18.0 and 30.0 kg/m2

Main Exclusion Criteria:

* History of any clinically-relevant gastrointestinal, renal, hepatic, bronchopulmonary, neurological, psychiatric, cardiovascular, endocrine, haematologic, neuromuscular or allergic disease(s), metabolic disorder, cancer, cirrhosis, significant acute infection, local infection within 2 weeks of dose administration,
* ECG: any history of clinically-significant ECG abnormalities, an uninterpretable ECG, or any of ECG abnormalities, unless considered not significant by the Investigator
* Abnormalities in clinical chemical, haematological, or coagulation variables considered medically relevant by the Investigator,
* Positive urine drug screen, positive breathalyzer for alcohol
* Positive results in any of the following virology tests: HIV-1 and -2 antibodies, HBsAg, and anti-hepatitis C virus antibody
* Positive SARS-CoV-2 antigen test
* Women who are pregnant or nursing,
* Donation or loss of over 500 mL of blood within sixty days prior to the first study drug administration,

Part C with co-administration of meropenem:

1. History of epilepsy (or known seizure disorder), brain lesions or other significant neurological disorders,
2. Known history of clinically-significant hypersensitivity or urticaria, or severe allergic reaction to β-lactam antibiotics,
3. History of Gilbert syndrome,
4. History of any severe antibiotic-associated superinfections,

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
Number and severity of Treatment Emergent Adverse Events (TEAE) to evaluate the safety and tolerability profile of single and multiple intravenous ascending doses of ANT3310 alone (Part A and B) and in combination with meropenem (Part C) | up to 11 days
  Percentage of subjects who experience at least one TEAE, including abnormalities in vital signs, physical examinations, laboratory safety tests and ECG, by seriousness, intensity, and relatedness

SECONDARY OUTCOMES:
Part A (SAD): Maximum Plasma Concentration (Cmax) of single i.v. ascending doses of ANT3310 alone | 24 hours
  Pharmacokinetic parameter of ANT3310 in plasma
Part A (SAD): Area under the concentration time curve (AUC) of single i.v. ascending doses of ANT3310 alone | 24 hours
  Pharmacokinetic parameter of ANT3310 in plasma
Part A (SAD): Time to maximum plasma concentration (Tmax) of single i.v. ascending doses of ANT3310 alone | 24 hours
  Pharmacokinetic parameter of ANT3310 in plasma
Part A (SAD): Half-time (t1/2) of single i.v. ascending doses of ANT3310 alone | 24 hours
  Pharmacokinetic parameter of ANT3310 in plasma
Part B (MAD): Maximum Plasma Concentration (Cmax) of multiple i.v. ascending doses of ANT3310 alone | Day 1, Day 7
  Pharmacokinetic parameter of ANT3310 in plasma
Part B (MAD): Area under the concentration time curve (AUC) of multiple i.v. ascending doses of ANT3310 alone | Day 1, Day 7
  Pharmacokinetic parameter of ANT3310 in plasma
Part B (MAD): Time to maximum plasma concentration (Tmax) of multiple i.v. ascending doses of ANT3310 alone | Day 1, Day 7
  Pharmacokinetic parameter of ANT3310 in plasma
Part C (DDI and combination): Maximum Plasma Concentration (Cmax) of a single i.v. dose of ANT3310 and meropenem | Day 1, Day 3, Day 5
  Pharmacokinetic parameter of ANT3310 and meropenem in plasma
Part C (DDI and combination): Area under the concentration time curve (AUC) of a single i.v. dose of ANT3310 and meropenem | Day 1, Day 3, Day 5
  Pharmacokinetic parameter of ANT3310 and meropenem in plasma
Part C (DDI and combination): Time to maximum plasma concentration (Tmax) of a single i.v. dose of ANT3310 and meropenem | Day 1, Day 3, Day 5
  Pharmacokinetic parameter of ANT3310 and meropenem in plasma
Part C (DDI and combination): Maximum Plasma Concentration (Cmax) of multiple i.v. dose of ANT3310 co-administered with meropenem | Day 11
  Pharmacokinetic parameter of ANT3310 and meropenem in plasma
Part C (DDI and combination): Area under the concentration time curve (AUC) of multiple i.v. dose of ANT3310 co-administered with meropenem | Day 11
  Pharmacokinetic parameter of ANT3310 and meropenem in plasma
Part C (DDI and combination): Time to maximum plasma concentration (Tmax) of multiple i.v. dose of ANT3310 co-administered with meropenem | Day 11
  Pharmacokinetic parameter of ANT3310 and meropenem in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Hays, MD, Principal Investigator — Biotrial
Locations (1):
- Biotrial, Rennes, France

IPD SHARING:
Plan to Share IPD: No